CLINICAL TRIAL: NCT00642564
Title: MIGRAINE AND HEADACHE IN EPILEPTIC PATIENTS
Brief Title: Study on Migraine and Headache in Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014668
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Headache; Migraine
MeSH Terms: conditions — Epilepsy; Headache; Migraine Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Observational study in Epileptic Patients

INTERVENTIONS:
Other: Observational study in Epileptic Patients — Observation study in Epileptic Patients with Migraine and Headache

SUMMARY:
The purpose of this study is to collect data from patients who are diagnosed with epilepsy and are followed up in epilepsy clinics.

DETAILED DESCRIPTION:
Headaches and epilepsy are chronic disorders with episodic manifestations characterized by recurrent attacks of nervous system dysfunction with a return to baseline between attacks. Although it is not uncommon that patients with epilepsy suffer from headaches, the relations between seizures and headaches is multi-factorial. Headaches may occur immediately before (preictal), during (ictal), or after (postictal) a seizure. In addition to seizure-associated headaches, patients often experience headaches that are not temporally related to seizures-interictal headaches. Moreover, epidemiological studies indicate an association of migraine and epilepsy with an increased prevalence of migraine in patients with epilepsy. Up to now, there is still limited information about the relationship between the frequency of seizure attacks and headache occurrences. Thus, we purpose this study to investigate the incidence of headaches, to explore the relationship between seizure attacks and headache occurrences, to classify the headache, and to document the frequency, characteristics, and effects of migraine and headaches among patients with epilepsy. This study is a multi-centre survey to collect data from patients who are diagnosed with epilepsy and are followed up in epilepsy clinics. Patients can only participate in this study after signing and dating the inform consents. There are two stages of this study: Stage I: On enrollment, data on demographic characteristics, epilepsy profile, seizure frequencies, and epilepsy treatment would be obtained. Body weight and height would be measured. Information of prior headache occurrences and their relationships with seizures would also be collected. Stage II: Patients enrolled into this study will be divided into three group: patients who are seizure free for past 6 months, patients with > 1 attack every month within past 6 months, and other patients. Participants of each group will be enrolled into Stage II for 24-week follow-up. Information of seizure attacks, headache occurrences, and treatment will be collected. This is an observational study and no study drug is administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with epilepsy
* Patients or parent(s)/caregiver(s) have signed and dated an informed consent.

Exclusion Criteria:

* Patients who have non-epileptic events in addition to epilepsy, such as pseudoseizures or an acute symptomatic cause of seizures (e.g., a metabolic disturbance, toxic exposure, active CNS infection)
* Patients with progressive or degenerative neurological disorder
* Patients with an active malignancy
* Patients or parents/caregivers with known or suspected psychotic disease, mental retardation, or any mental situation which may cause the concern to properly complete this survey.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll patients with diagnosis of epilepsy and age should be equal or more than 7 years old.
Sampling Method: Probability Sample
Enrollment: 955 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and the frequencies of migraines and other types of headache among patients with epilepsy, and to explore the relationship between seizure frequencies and headache occurrences | Participants of each group will be enrolled for 24-week follow-up.

SECONDARY OUTCOMES:
A decreased number of seizure symptoms as noted by the improved score on the 10-point Visual Analog Scale | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd